CLINICAL TRIAL: NCT04098575
Title: Treatment of T2DM Patients in Germany Receiving Empagliflozin: A Retrospective RWE Study Description of Treatment and Population Characteristics of Type 2 Diabetic Patients in Germany Receiving Empagliflozin: A Retrospective Real-World Evidence (RWE) Study Based on German Registries DPV&DIVE
Brief Title: A Study Based on Data From German Registries That Looks at Characteristics of People Who Take the Medicine Empagliflozin for Type 2 Diabetes
Acronym: EDCOS
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1245-0198
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Results first posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Patients receiving Empagliflozin until mid Sep 2015: Patients receiving Empagliflozin before the EMPA-REG-OUTCOME study was published time until mid-Sept. 2015; Cohort 1
  Interventions: Drug: Empagliflozin
- Patients receiving Empagliflozin until CV Label Change time: Patients receiving Empagliflozin starting from the EMPA-REG-OUTCOME study being published until CV Label Change time from mid-Sept. 2015-mid-Jan. 2017; Cohort 2
  Interventions: Drug: Empagliflozin
- Patients receiving Empagliflozin until last available data cut: Patients receiving Empagliflozin starting from mid-Jan. 2017 until last; Cohort 3
  Interventions: Drug: Empagliflozin

INTERVENTIONS:
Drug: Empagliflozin — drug

SUMMARY:
Description of the real-life treatment of adult patients with type-2 diabetes mellitus (T2DM) receiving Empagliflozin, comparing the characteristics of patients starting Empagliflozin in three time intervals

ELIGIBILITY:
Inclusion Criteria:

* At least two outpatient T2DM diagnoses (ICD E11.-) in two different quarters and/or at least one inpatient T2DM diagnosis (ICD E11)
* At least one prescription of an empagliflozin-containing antidiabetic drug: Jardiance® (Empagliflozin, ATC A10BK03, former A10BX12) or Synjardy® (Empagliflozin/ Met¬for¬min, ATC A10BD20)

Exclusion Criteria:

* Any diagnosis of T1DM

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Diabetes Mellitus, Type 2, treated with Empagliflozin
Sampling Method: Non-Probability Sample
Enrollment: 9571 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Diabetes Agenda 2010 GmbH, Mahlow, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. Studies in products where Boehringer Ingelheim is not the license holder
  2. Studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials
  3. Studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  Requestors can use the following link http://trials.boehringer-ingelheim.com/

REFERENCES:
- See also: Related Info — http://mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A retrospective real-world evidence study based on existing data to describe the treatment and population characteristics of patients with type-2 diabetes mellitus (T2DM) receiving empagliflozin in thee time intervals.
Pre-assignment Details: All patients were screened for eligibility to participate in the trial. Only patients that met all the inclusion and none of the exclusion criteria were included in the trial.
Groups:
- Early Users: Patients Receiving Empagliflozin Until Mid-September 2015: Data from two german patient registries (Diabetes-Patienten-Verlaufs-Dokumentations (DPV) and Diabetes Versorgungs-Evaluation (DIVE)) on patients with type 2 diabetes mellitus (T2DM), registered between 2014 and 2019, receiving empagliflozin were used. Cohort 1 (early users) included only patients who received empagliflozin before the EMPA-REG OUTCOME study publication in mid-September 2015.
- Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017: Data from two german patient registries (Diabetes-Patienten-Verlaufs-Dokumentations (DPV) and Diabetes Versorgungs-Evaluation (DIVE)) on patients with T2DM, registered between 2014 and 2019, receiving empagliflozin were used. Cohort 2 (intermediate users) included only patients who started empagliflozin after the EMPA-REG OUTCOME study publication (mid-September 2015), but before the European Medicines Agency label change (mid-January 2017).
- Late Users: Patients Receiving Empagliflozin After Mid-January 2017: Data from two german patient registries (Diabetes-Patienten-Verlaufs-Dokumentations (DPV) and Diabetes Versorgungs-Evaluation (DIVE)) on patients with T2DM, registered between 2014 and 2019, receiving empagliflozin were used. Cohort 3 (late users) included only patients who started empagliflozin after mid-January 2017 until last available data cut in September 2019.
Period: Overall Study
Arm/Group | Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 | Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 | Late Users: Patients Receiving Empagliflozin After Mid-January 2017
Started | 505 | 2961 | 6105
Completed | 505 | 2961 | 6105
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients from the two largest German registries (Diabetes-Patienten-Verlaufs-Dokumentation and Diabetes Versorgungs-Evaluation) with Type-2 Diabetes Mellitus and with empagliflozin treatment were included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 | Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 | Late Users: Patients Receiving Empagliflozin After Mid-January 2017 | Total
Number analyzed (Participants) | 505 | 2961 | 6105 | 9571
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.2 (11.3) | 61.2 (11.5) | 63.2 (11.4) | 62.4 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 248 | 1131 | 2045 | 3424
  Male | 257 | 1830 | 4060 | 6147
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Previous Occurence of Cardiovascular Comorbidities
Description: Percentage of patients with previous occurence of cardiovascular (CV) comorbidities, including myocardial infarction, stroke, coronary artery disease, peripheral arterial disease, congestive heart failure.
Time Frame: At baseline.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 | Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 | Late Users: Patients Receiving Empagliflozin After Mid-January 2017
Number analyzed (Participants) | 505 | 2961 | 6105
Percentage of participants | 20.4 | 21.6 | 26.4
Statistical Analysis 1: Comparison: Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 vs Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 vs Late Users: Patients Receiving Empagliflozin After Mid-January 2017; Test type: Other; p < 0.001, Chi-squared

2. Primary Outcome: Percentage of Participants With Previous Occurence of Other Typical Diabetes Complications
Description: Percentage of participants with previous occurence of other typical diabetes complications, including, Neuropathy, Nephropathy, Chronic Kidney Disease, Microalbuminuria, Macroalbuminuria, estimated glomerular filtration rate (eGFR), diabetic foot syndrome, retinopathy (background and proliferative).
Time Frame: At baseline.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 | Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 | Late Users: Patients Receiving Empagliflozin After Mid-January 2017
Number analyzed (Participants) | 505 | 2961 | 6105
Percentage of participants | 59.6 | 57.6 | 59.8
Statistical Analysis 1: Comparison: Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 vs Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 vs Late Users: Patients Receiving Empagliflozin After Mid-January 2017; Test type: Other; p = 0.835, Chi-squared

3. Primary Outcome: Percentage of Participants With Antidiabetic and Cardiovascular Co-medication
Description: Percentage of participants with antidiabetic and cardiovascular co-medication, including lipid-lowering agents, other antihypertensives, antiplatelets and anticoagulants.
Time Frame: At baseline.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 | Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 | Late Users: Patients Receiving Empagliflozin After Mid-January 2017
Number analyzed (Participants) | 505 | 2961 | 6105
Percentage of participants
  Antihypertensive drugs | 45.4 | 49.5 | 59.8
  Lipid-lowering agents | 28.3 | 36.4 | 46.0
  Antplatelet, anticoagulant drugs | 11.7 | 17.4 | 25.3
  Glucose-lowering therapies | 80.2 | 83.1 | 90.6
Statistical Analysis 1: Comparison: Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 vs Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 vs Late Users: Patients Receiving Empagliflozin After Mid-January 2017; Antihypertensive drugs; Test type: Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 vs Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 vs Late Users: Patients Receiving Empagliflozin After Mid-January 2017; Lipid-lowering agents; Test type: Other; p < 0.001, Chi-squared
Statistical Analysis 3: Comparison: Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 vs Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 vs Late Users: Patients Receiving Empagliflozin After Mid-January 2017; Antiplatelet, anticoagulant drugs; Test type: Other; p < 0.001, Chi-squared
Statistical Analysis 4: Comparison: Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 vs Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 vs Late Users: Patients Receiving Empagliflozin After Mid-January 2017; Glucose-lowering therapies; Test type: Other; p < 0.001, Chi-squared

4. Secondary Outcome: Percentage of Participants by Age Category
Description: Percentage of participants by age category; younger than 65 (< 65), from 65 to 74 (65 ≤ 75) , from 75 to 80 (75 - 80) , older than 80 (> 80).
Time Frame: At baseline.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 | Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 | Late Users: Patients Receiving Empagliflozin After Mid-January 2017
Number analyzed (Participants) | 505 | 2961 | 6105
Percentage of participants
  < 65 | 71.1 | 60.8 | 54.4
  65 ≤ 75 | 20.0 | 27.4 | 28.9
  75 - 80 | 6.5 | 8.3 | 11.3
  > 80 | 2.4 | 3.6 | 5.4
Statistical Analysis 1: Comparison: Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 vs Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 vs Late Users: Patients Receiving Empagliflozin After Mid-January 2017; Group: < 65; Test type: Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 vs Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 vs Late Users: Patients Receiving Empagliflozin After Mid-January 2017; Group: 65 ≤ 75; Test type: Other; p = 0.001, Chi-squared
Statistical Analysis 3: Comparison: Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 vs Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 vs Late Users: Patients Receiving Empagliflozin After Mid-January 2017; Group: 75 - 80; Test type: Other; p < 0.001, Chi-squared
Statistical Analysis 4: Comparison: Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 vs Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 vs Late Users: Patients Receiving Empagliflozin After Mid-January 2017; Group: > 80; Test type: Other; p < 0.002, Chi-squared

5. Secondary Outcome: Percentage of Male Participants
Description: The percentage of male participants is reported.
Time Frame: At baseline.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 | Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 | Late Users: Patients Receiving Empagliflozin After Mid-January 2017
Number analyzed (Participants) | 505 | 2961 | 6105
Percentage of participants | 50.9 | 61.8 | 66.5
Statistical Analysis 1: Comparison: Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 vs Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 vs Late Users: Patients Receiving Empagliflozin After Mid-January 2017; Test type: Other; p < 0.001, Chi-squared

6. Secondary Outcome: Weight of Participants
Description: Weight of participants.
Time Frame: At baseline.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 | Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 | Late Users: Patients Receiving Empagliflozin After Mid-January 2017
Number analyzed (Participants) | 505 | 2961 | 6105
Kilogram (kg) | 103.2 (21.4) | 100.3 (23.1) | 97.3 (21.7)
Statistical Analysis 1: Comparison: Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 vs Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 vs Late Users: Patients Receiving Empagliflozin After Mid-January 2017; Test type: Other; p < 0.001, Wilcoxon rank sum test

7. Secondary Outcome: Height of Participants
Description: Height of participants.
Time Frame: At baseline.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Centimeter (cm)
Arm/Group | Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 | Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 | Late Users: Patients Receiving Empagliflozin After Mid-January 2017
Number analyzed (Participants) | 505 | 2961 | 6105
Centimeter (cm) | 170.5 (9.5) | 171.8 (9.9) | 172.3 (9.6)
Statistical Analysis 1: Comparison: Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 vs Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 vs Late Users: Patients Receiving Empagliflozin After Mid-January 2017; Test type: Other; p < 0.001, Wilcoxon rank sum test

8. Secondary Outcome: Glycated Hemoglobin (HbA1c)
Description: Glycated hemoglobin (HbA1c).
Time Frame: At baseline.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: nanomol/mol
Arm/Group | Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 | Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 | Late Users: Patients Receiving Empagliflozin After Mid-January 2017
Number analyzed (Participants) | 505 | 2961 | 6105
nanomol/mol | 65.7 (18.4) | 66.6 (18.7) | 67.8 (20.4)
Statistical Analysis 1: Comparison: Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 vs Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 vs Late Users: Patients Receiving Empagliflozin After Mid-January 2017; Test type: Other; p = 0.475, Wilcoxon rank sum test

9. Secondary Outcome: Duration of Diabetes
Description: Duration of diabetes (time since diagnosis).
Time Frame: At baseline.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 | Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 | Late Users: Patients Receiving Empagliflozin After Mid-January 2017
Number analyzed (Participants) | 505 | 2961 | 6105
Years | 10.7 (7.8) | 10.8 (8.2) | 11.2 (8.5)
Statistical Analysis 1: Comparison: Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 vs Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 vs Late Users: Patients Receiving Empagliflozin After Mid-January 2017; Test type: Other; p = 0.475, Wilcoxon rank sum test

10. Secondary Outcome: Percentage of Participants With Previous Glucose-lowering Treatment
Description: Percentage of participants with glucose-lowering treatment prior to empagliflozin initiation.
Time Frame: At baseline.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 | Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 | Late Users: Patients Receiving Empagliflozin After Mid-January 2017
Number analyzed (Participants) | 505 | 2961 | 6105
Percentage of participants
  Insulin | 34.3 | 37.2 | 49.9
  Metformin | 60.8 | 59.7 | 68.6
  Acarbose | 1.0 | 0.9 | 0.4
  Sulfonylurea | 9.3 | 6.8 | 5.0
  Dipeptidyl peptidase-4 (DPP-4) inhibitors | 25.2 | 31.1 | 31.8
  Glucagon-like peptide-1 (GLP-1) agonists | 12.1 | 12.2 | 13.9
  Sodium-glucose transport protein-2 (SGLT2) inhibitors other than empagliflozin | 7.9 | 2.3 | 2.7
Statistical Analysis 1: Comparison: Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 vs Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 vs Late Users: Patients Receiving Empagliflozin After Mid-January 2017; Insulin; Test type: Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 vs Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 vs Late Users: Patients Receiving Empagliflozin After Mid-January 2017; Metformin; Test type: Other; p < 0.001, Chi-squared
Statistical Analysis 3: Comparison: Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 vs Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 vs Late Users: Patients Receiving Empagliflozin After Mid-January 2017; Acarbose; Test type: Other; p = 0.157, Chi-squared
Statistical Analysis 4: Comparison: Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 vs Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 vs Late Users: Patients Receiving Empagliflozin After Mid-January 2017; Sulfonylurea; Test type: Other; p < 0.001, Chi-squared
Statistical Analysis 5: Comparison: Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 vs Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 vs Late Users: Patients Receiving Empagliflozin After Mid-January 2017; Dipeptidyl peptidase-4 (DPP-4) inhibitors; Test type: Other; p = 0.071, Chi-squared
Statistical Analysis 6: Comparison: Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 vs Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 vs Late Users: Patients Receiving Empagliflozin After Mid-January 2017; Glucagon-like peptide-1 (GLP-1) agonists; Test type: Other; p = 0.317, Chi-squared
Statistical Analysis 7: Comparison: Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 vs Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 vs Late Users: Patients Receiving Empagliflozin After Mid-January 2017; Sodium-glucose transport protein-2 (SGLT2) inhibitors other than empagliflozin; Test type: Other; p < 0.001, Chi-squared

11. Secondary Outcome: Percentage of Patients Participated in Disease Management Programme (DMP) Type 2 Diabetes
Description: Percentage of patients participated in Disease Management Programme (DMP) Type 2 Diabetes.
Time Frame: At baseline.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 | Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 | Late Users: Patients Receiving Empagliflozin After Mid-January 2017
Number analyzed (Participants) | 505 | 2961 | 6105
Percentage of participants | 53.5 | 48.6 | 31.8
Statistical Analysis 1: Comparison: Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 vs Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 vs Late Users: Patients Receiving Empagliflozin After Mid-January 2017; Test type: Other; p < 0.002, Chi-squared

12. Secondary Outcome: Number of Participants With Hospitalizations
Description: Number of participants with hospitalizations.
Time Frame: At baseline.
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 | Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 | Late Users: Patients Receiving Empagliflozin After Mid-January 2017
Number analyzed (Participants) | 505 | 2961 | 6105
Participants | NA — Data on hospitalizations were not included on the registries, thus no data were available for analysis. | NA — Data on hospitalizations were not included on the registries, thus no data were available for analysis. | NA — Data on hospitalizations were not included on the registries, thus no data were available for analysis.

13. Secondary Outcome: Dosage of Empagliflozin
Description: Dosage of empagliflozin. Number of patients on 10 milligram versus patients on 25 milligram empagliflozin.
Time Frame: At baseline.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 | Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 | Late Users: Patients Receiving Empagliflozin After Mid-January 2017
Number analyzed (Participants) | 505 | 2961 | 6105
Participants
  10 milligram of empagliflozin | NA — Data on dosage of empagliflozin were not included on the registries, thus no data were available for analysis. | NA — Data on dosage of empagliflozin were not included on the registries, thus no data were available for analysis. | NA — Data on dosage of empagliflozin were not included on the registries, thus no data were available for analysis.
  25 milligram of empagliflozin | NA — Data on dosage of empagliflozin were not included on the registries, thus no data were available for analysis. | NA — Data on dosage of empagliflozin were not included on the registries, thus no data were available for analysis. | NA — Data on dosage of empagliflozin were not included on the registries, thus no data were available for analysis.

14. Secondary Outcome: Fasting Plasma Glucose (FPG)
Description: Fasting plasma glucose (FPG).
Time Frame: At baseline.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Milligram / deciliter
Arm/Group | Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 | Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 | Late Users: Patients Receiving Empagliflozin After Mid-January 2017
Number analyzed (Participants) | 505 | 2961 | 6105
Milligram / deciliter | 186.0 (85.6) | 182.3 (76.5) | 181.1 (78.5)
Statistical Analysis 1: Comparison: Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 vs Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 vs Late Users: Patients Receiving Empagliflozin After Mid-January 2017; Test type: Other; p = 1.000, Wilcoxon rank sum test

ADVERSE EVENTS:
Description: As this is a non-interventional study with secondary use of data retrieved from a US health claims database, safety monitoring and safety reporting on an individual case level is not applicable. "0" total Number of Participants at Risk means "All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed".
Arm/Group | Early Users: Patients Receiving Empagliflozin Until Mid-September 2015 | Intermediate Users: Patients Receiving Empagliflozin From Mid-September 2015 to Mid-January 2017 | Late Users: Patients Receiving Empagliflozin After Mid-January 2017
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The main limitation of the study is that patients were recruited from specialized centers that were participating in diabetes registries, which could bias the results toward patients requiring specialist care. The cross-sectional nature of the study precludes the identification of causal links between findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-16): https://cdn.clinicaltrials.gov/large-docs/75/NCT04098575/Prot_SAP_000.pdf